CLINICAL TRIAL: NCT04848610
Title: Evaluation of The Factors That Affect The Infection Of Covid-19 In Turkish Society
Brief Title: The Factors That Affect the Infection of COVID-19
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulbeyaz Can, Prof.Dr., Istanbul University - Cerrahpasa
Other Study IDs: Covid-19 Infection
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: COVID-19 Infection
Keywords: COVID-19; risk factor; symptoms; protective measures
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The number of new Coronavirus-2019 (Covid-19) cases is increasing day by day despite the warnings "Stay at home! Wear a mask! Keep social distance!". The aim of this descriptive study is to determine the risk factors that affect the Covid-19 infection in Turkey.

The online link of the form created on Google forms was sent to the participants' phones between 18.10.2020 and 18.11.2020.

DETAILED DESCRIPTION:
The number of new Coronavirus-2019 (Covid-19) cases is increasing day by day despite the warnings "Stay at home! Wear a mask! Keep social distance!". The aim of this descriptive study is to determine the risk factors that affect the Covid-19 infection in Turkey.

The majority of the lands within the Republic of Turkey cover Anatolia, while a minor part covers Thrace, the southeast extension of the Balkan Peninsula. The population of Turkey is 83,154,997. Based on the natural, human and financial characteristics, the country consists of seven regions: Mediterranean, Eastern Anatolia, Aegean, Southeastern Anatolia, Central Anatolia, Marmara, and Black Sea. The majority of the population lives in the Marmara Region. The online link of the form created on Google forms was sent to the participants' phones between 18.10.2020 and 18.11.2020 and participants' informed consent was obtained.

A 43-item questionnaire form which had two sections and was prepared by the researcher in line with the literature was used in data collection. The first section questioned participants' personal characteristics (first letters of participants' names and surnames, date of birth, profession, employment status, risk of Covid-19 infection, family type, etc.), while the second section questioned the practices of following 14 rules declared by the Turkish Ministry of Health to prevent the Covid-19 pandemic (using a mask, observing the hand hygiene and social distance, etc.) and whether participants were diagnosed with Covid-19. Identity details that could help identify the participants were not questioned.

ELIGIBILITY:
Inclusion Criteria:

* Being over the age of 18
* Be in good mental and mental health
* To be able to read and write

Exclusion Criteria:

* Being under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The majority of the lands within the Republic of Turkey cover Anatolia, while a minor part covers Thrace, the southeast extension of the Balkan Peninsula. The population of Turkey is 83,154,997. Based on the natural, human and financial characteristics, the country consists of seven regions: Mediterranean, Eastern Anatolia, Aegean, Southeastern Anatolia, Central Anatolia, Marmara, and Black Sea. The majority of the population lives in the Marmara Region. Many people from seven regions of Turkey were invited to participate in the study, only 1264 individuals participated. The data of 1104 people who agreed to participate and completed the assessment form thoroughly were included. Data of 160 were excluded owing to answering certain items twice.
Sampling Method: Non-Probability Sample
Enrollment: 1104 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Risk factors affecting the infection of Covid-19 in Turkish society | Last 6 month
  Risk factors for Covid-19 infection

SECONDARY OUTCOMES:
Difference between the protective measures taken from Covid-19 cases and healthy people | Last 6 month
  Protective measures taken during the Covid-19 Pandemic

CONTACTS AND LOCATIONS:
Overall Officials: Gulbeyaz CAN, Prof., Principal Investigator — IUC Florence Nıghtingale Nursing Faculty
Locations (1):
- Istanbul University-Cerrahpasa Florence Nightingale Nursing Faculty, Istanbul, Turkey (Türkiye)